CLINICAL TRIAL: NCT05335707
Title: Longitudinal Geriatric Assessment to Optimize Outcomes of Older Patients With Muscle-Invasive Bladder Cancer After Radical Cystectomy: A Pilot Trial
Brief Title: Longitudinal Geriatric Assessment to Optimize Outcomes of Older Patients With Muscle-Invasive Bladder Cancer After Radical Cystectomy
Status: Withdrawn | Type: Observational
Why Stopped: Study funds ended on 7/31/2023
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Wulff-Burchfield, MD, Assistant Professor, University of Kansas Medical Center
Other Study IDs: IIT-2021-GerioncBladder
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single arm pilot study will evaluate the feasibility and acceptability for perioperative Comprehensive Geriatric Assessment (CGA) and CGA-directed supportive and restorative care for patients with muscle-invasive bladder cancer who are planned to undergo preoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males and females age ≥ 65 years
* Diagnosis/disease status
* Histologically proven muscle-invasive bladder cancer (MIBC) without metastatic disease.
* Patients planning to undergo neoadjuvant chemotherapy and radical cystectomy for MIBC.
* Treatment with investigational systemic therapy is permitted if participants will be receiving chemotherapy as part of their treatment plan

Exclusion Criteria:

* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Any other known invasive malignancy within previous 2 years with the following EXCEPT: low grade prostate cancer on active surveillance, chronic lymphocytic leukemia CLL on surveillance / observation, non-melanoma skin cancers

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 and older with biopsy-proven muscle-invasive bladder cancer planned for neoadjuvant chemotherapy and radical cystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Develop a geriatric oncology assessment clinic and workflows | 12 months
  Develop a geriatric oncology assessment clinic and workflows for the University of Kansas Health System, including University of Kansas Cancer Center St. Francis and Great Bend practices.

SECONDARY OUTCOMES:
Test feasibility, acceptability, and preliminary impact | 12 months
  Test feasibility, acceptability, and preliminary impact of the Comprehensive Geriatric Assessment (CGA) and CGA-directed care.
  Note: The results of the CGA will be used by clinicians to guide patients' medical care.